CLINICAL TRIAL: NCT02522559
Title: Using Herbs and Spices to Increase Children's Acceptance and Intake of Vegetables in School Lunches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Director, Metabolic Kitchen & Children's Eating Behavior Lab, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Spiceinschool01; Spices (Other: McCormick Science Institute)
Record Dates: First submitted 2015-04-06; First posted 2015-08-13 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spice Intervention (Experimental): Spice intervention: Student-approved vegetable recipes will be served in the school cafeteria.
  Interventions: Other: Spice Intervention

INTERVENTIONS:
Other: Spice Intervention — Spice Intervention:Novel herb and spice blends will be used in cafeteria recipes.

SUMMARY:
Herbs and spices offer one potential solution to the recent decline in children taking school lunch because they can increase the palatability of foods without adding salt and fat. However, there is currently limited evidence on how to successfully integrate herbs and spices into the school lunch menu. Developing evidence-based methods to teach school cafeteria workers to prepare healthy and tasty vegetable dishes with the addition of herbs and spices is a research priority. The investigators hypothesize that herbs and spices can be used to increase acceptance, intake, and participation in the school lunch program among 6th - 12th grade students from Central Pennsylvania.

DETAILED DESCRIPTION:
What this study will add to the literature: Herbs and spices offer one potential solution to the recent decline in children taking school lunch because they can increase the palatability of foods without adding salt and fat. However, there is currently limited evidence on how to successfully integrate herbs and spices into the school lunch menu. Developing evidence-based methods to teach school cafeteria workers to prepare healthy and tasty vegetable dishes with the addition of herbs and spices is a research priority. This research will provide evidence that herbs and spices can be used to increase acceptance, intake, and participation in the school lunch program among 6th - 12th grade students from Central Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

* Student in Bald Eagle Area Middle/High School
* Parents of students in Bald Eagle Area Middle/High School
* School Food Service Employees at the Bald Eagle Area Middle/High School

Exclusion Criteria:

* Students/children who have food allergies to herb/spice blend ingredients.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Surveys defining barriers to vegetable consumption at Bald Eagle Area Middle/High School | Baseline
  Conduct surveys of students, parents and food service experts to gather information describing ways to increase vegetable intake at Bald Eagle Area Middle/High School
Taste tests to quantify the change in liking of vegetable recipes | Baseline and after recipe development (approximately 10 months). Prior to intervention.
  Student's liking of vegetables prepared with herbs/spices will be assessed during the taste tests by setting up sensory panels in their culinary and consumer education classes. Participating students will rate liking and will provide written feedback to inform recipe development.
Change in vegetable plate waste | Baseline, Intervention and Follow-up (1 and 6 months)
  Weight of vegetable disappearance from the school cafeteria, minus waste weight, in kg.

SECONDARY OUTCOMES:
School lunch program participation | Baseline, Intervention and Followup (1 and 6 months)
  Percentage of children who are participating in the school lunch program will be assessed the school years prior to and immediately after the intervention
Post-meal comment cards | Baseline, Intervention and Followup (1 and 6 months)
  Student's will rate satisfaction with the school lunches by completing anonymous, post-meal comment cards during the baseline, intervention, and follow-up phases.

OTHER OUTCOMES:
Age Covariate | Baseline
  We plan to assess age to see if this covariate influences a student's response to the survey.
Weight Status Covariate | Baseline
  We plan to assess weight status to see if this covariate influences a student's response to the survey.
Parental Feeding Practices Covariate | Baseline
  We plan to assess if this covariate influences a student's response to the survey.
Parental Education Covariate | Baseline
  We plan to assess if this covariate influences a student's response to the survey.
Family Culture Covariate | Baseline
  We plan to assess if this covariate influences a student's response to the survey.
Family Intake of Herbs/Spices at Home Covariate | Baseline
  We plan to assess if this covariate influences a student's response to the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L. Keller, PhD, Principal Investigator — Penn State University
Locations (1):
- Bald Eagle Middle/High School, Wingate, Pennsylvania, United States